CLINICAL TRIAL: NCT04033965
Title: Tumor Mutational Patterns and Infiltrating Lymphocyte Density in Young and Old Patients With Breast Cancer
Brief Title: Corellation of Mutations, TILs and Age in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Principal Investigator, Manto Nikolaidi, Medical Oncologist, Hellenic Cooperative Oncology Group
Other Study IDs: HE10/mut
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — formalin-fixed paraffin-embedded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women <35 with early breast cancer
  Interventions: Genetic: Corellation of Mutations, TILs and Age in Breast Cancer
- women>65 years old with early breast cancer
  Interventions: Genetic: Corellation of Mutations, TILs and Age in Breast Cancer

INTERVENTIONS:
Genetic: Corellation of Mutations, TILs and Age in Breast Cancer

SUMMARY:
Age may pertain to different tumor genotype characteristics which may interfere with treatment efficacy and prognosis. The investigators investigated the distribution and prognostic effect of mutations (mut) and tumor infiltrating lymphocyte (TILs) in young and elderly early breast cancer patients (pts).

ELIGIBILITY:
Inclusion Criteria:

* women with early breast cancer <35 years old or >65 years old

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women with early breast cancer <35 years old or >65 years old
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 1997-09-03 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2010-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the prevalence of gene mutations in women <=35 years old with early breast cancer. | Up to 13 years
Assessment of the prevalence of gene mutations in women >65years old with early breast cancer. | Up to 13 years
Evaluation of Tumor Infiltrating Lymphocytes (TILs) density using descriptive statistics in women <=35 years old with early breast cancer. | Up to 13 years
Evaluation of Tumor Infiltrating Lymphocytes (TILs) density using descriptive statistics in women >65 years old with early breast cancer. | Up to 13 years
Evaluation of the prognostic effect of gene mutations and Tumor Infiltrating Lymphocytes with respect to Overall Survival in women <=35 years old with early breast cancer | Up to 13 years
Evaluation of the prognostic effect of gene mutations and Tumor Infiltrating Lymphocytes with respect to Overall Survival in women >65 years old with early breast cancer. | Up to 13 years

CONTACTS AND LOCATIONS:
Overall Officials: Adamantia Nikolaidi, MD, Principal Investigator — Oncology Department, MITERA Hospital

REFERENCES:
- [Background] Gnerlich JL, Deshpande AD, Jeffe DB, Sweet A, White N, Margenthaler JA. Elevated breast cancer mortality in women younger than age 40 years compared with older women is attributed to poorer survival in early-stage disease. J Am Coll Surg. 2009 Mar;208(3):341-7. doi: 10.1016/j.jamcollsurg.2008.12.001. Epub 2009 Jan 21. PMID 19317994
- [Background] Stickeler E. Prognostic and Predictive Markers for Treatment Decisions in Early Breast Cancer. Breast Care (Basel). 2011;6(3):193-198. doi: 10.1159/000329471. Epub 2011 Jun 14. PMID 21779224
- [Background] Bonnier P, Romain S, Charpin C, Lejeune C, Tubiana N, Martin PM, Piana L. Age as a prognostic factor in breast cancer: relationship to pathologic and biologic features. Int J Cancer. 1995 Jul 17;62(2):138-44. doi: 10.1002/ijc.2910620205. PMID 7622286
- [Background] Sweeney C, Blair CK, Anderson KE, Lazovich D, Folsom AR. Risk factors for breast cancer in elderly women. Am J Epidemiol. 2004 Nov 1;160(9):868-75. doi: 10.1093/aje/kwh276. PMID 15496539
- [Background] Gomez-Flores-Ramos L, Castro-Sanchez A, Pena-Curiel O, Mohar-Betancourt A. Molecular Biology In Young Women With Breast Cancer: From Tumor Gene Expression To DNA Mutations. Rev Invest Clin. 2017 Jul-Aug;69(4):181-192. doi: 10.24875/ric.17002225. PMID 28776603
- [Background] Azim HA Jr, Partridge AH. Biology of breast cancer in young women. Breast Cancer Res. 2014 Aug 27;16(4):427. doi: 10.1186/s13058-014-0427-5. PMID 25436920
- [Background] Aebi S, Gelber S, Castiglione-Gertsch M, Gelber RD, Collins J, Thurlimann B, Rudenstam CM, Lindtner J, Crivellari D, Cortes-Funes H, Simoncini E, Werner ID, Coates AS, Goldhirsch A. Is chemotherapy alone adequate for young women with oestrogen-receptor-positive breast cancer? Lancet. 2000 May 27;355(9218):1869-74. doi: 10.1016/s0140-6736(00)02292-3. PMID 10866443
- [Background] Arriagada R, Le MG, Dunant A, Tubiana M, Contesso G. Twenty-five years of follow-up in patients with operable breast carcinoma: correlation between clinicopathologic factors and the risk of death in each 5-year period. Cancer. 2006 Feb 15;106(4):743-50. doi: 10.1002/cncr.21659. PMID 16411216
- [Background] Goldhirsch A, Gelber RD, Yothers G, Gray RJ, Green S, Bryant J, Gelber S, Castiglione-Gertsch M, Coates AS. Adjuvant therapy for very young women with breast cancer: need for tailored treatments. J Natl Cancer Inst Monogr. 2001;(30):44-51. doi: 10.1093/oxfordjournals.jncimonographs.a003459. PMID 11773291
- [Background] Kroman N, Jensen MB, Wohlfahrt J, Mouridsen HT, Andersen PK, Melbye M. Factors influencing the effect of age on prognosis in breast cancer: population based study. BMJ. 2000 Feb 19;320(7233):474-8. doi: 10.1136/bmj.320.7233.474. PMID 10678859
- [Background] Encinas G, Sabelnykova VY, de Lyra EC, Hirata Katayama ML, Maistro S, de Vasconcellos Valle PWM, de Lima Pereira GF, Rodrigues LM, de Menezes Pacheco Serio PA, de Gouvea ACRC, Geyer FC, Basso RA, Pasini FS, Del Pilar Esteves Diz M, Brentani MM, Guedes Sampaio Goes JC, Chammas R, Boutros PC, Koike Folgueira MAA. Somatic mutations in early onset luminal breast cancer. Oncotarget. 2018 Apr 27;9(32):22460-22479. doi: 10.18632/oncotarget.25123. eCollection 2018 Apr 27. PMID 29854292
- [Background] Kotoula V, Karavasilis V, Zagouri F, Kouvatseas G, Giannoulatou E, Gogas H, Lakis S, Pentheroudakis G, Bobos M, Papadopoulou K, Tsolaki E, Pectasides D, Lazaridis G, Koutras A, Aravantinos G, Christodoulou C, Papakostas P, Markopoulos C, Zografos G, Papandreou C, Fountzilas G. Effects of TP53 and PIK3CA mutations in early breast cancer: a matter of co-mutation and tumor-infiltrating lymphocytes. Breast Cancer Res Treat. 2016 Jul;158(2):307-21. doi: 10.1007/s10549-016-3883-z. Epub 2016 Jul 1. PMID 27369359
- [Background] Papaxoinis G, Kotoula V, Alexopoulou Z, Kalogeras KT, Zagouri F, Timotheadou E, Gogas H, Pentheroudakis G, Christodoulou C, Koutras A, Bafaloukos D, Aravantinos G, Papakostas P, Charalambous E, Papadopoulou K, Varthalitis I, Efstratiou I, Zaramboukas T, Patsea H, Scopa CD, Skondra M, Kosmidis P, Pectasides D, Fountzilas G. Significance of PIK3CA Mutations in Patients with Early Breast Cancer Treated with Adjuvant Chemotherapy: A Hellenic Cooperative Oncology Group (HeCOG) Study. PLoS One. 2015 Oct 9;10(10):e0140293. doi: 10.1371/journal.pone.0140293. eCollection 2015. PMID 26452060
- [Background] Kotoula V, Chatzopoulos K, Lakis S, Alexopoulou Z, Timotheadou E, Zagouri F, Pentheroudakis G, Gogas H, Galani E, Efstratiou I, Zaramboukas T, Koutras A, Aravantinos G, Samantas E, Psyrri A, Kourea H, Bobos M, Papakostas P, Kosmidis P, Pectasides D, Fountzilas G. Tumors with high-density tumor infiltrating lymphocytes constitute a favorable entity in breast cancer: a pooled analysis of four prospective adjuvant trials. Oncotarget. 2016 Jan 26;7(4):5074-87. doi: 10.18632/oncotarget.6231. PMID 26506242
- [Background] Kotoula V, Lyberopoulou A, Papadopoulou K, Charalambous E, Alexopoulou Z, Gakou C, Lakis S, Tsolaki E, Lilakos K, Fountzilas G. Evaluation of two highly-multiplexed custom panels for massively parallel semiconductor sequencing on paraffin DNA. PLoS One. 2015 Jun 3;10(6):e0128818. doi: 10.1371/journal.pone.0128818. eCollection 2015. PMID 26039550
- [Background] Sun H, Yu G. New insights into the pathogenicity of non-synonymous variants through multi-level analysis. Sci Rep. 2019 Feb 7;9(1):1667. doi: 10.1038/s41598-018-38189-9. PMID 30733553
- [Background] Martincorena I, Raine KM, Gerstung M, Dawson KJ, Haase K, Van Loo P, Davies H, Stratton MR, Campbell PJ. Universal Patterns of Selection in Cancer and Somatic Tissues. Cell. 2017 Nov 16;171(5):1029-1041.e21. doi: 10.1016/j.cell.2017.09.042. Epub 2017 Oct 19. PMID 29056346
- [Background] Poggio F, Lambertini M, Bighin C, Conte B, Blondeaux E, D'Alonzo A, Dellepiane C, Boccardo F, Del Mastro L. Management of young women with early breast cancer. ESMO Open. 2018 Nov 14;3(Suppl 1):e000458. doi: 10.1136/esmoopen-2018-000458. eCollection 2018. PMID 30559981
- [Background] Cancer Genome Atlas Network. Comprehensive molecular portraits of human breast tumours. Nature. 2012 Oct 4;490(7418):61-70. doi: 10.1038/nature11412. Epub 2012 Sep 23. PMID 23000897
- [Background] Hobert JA, Eng C. PTEN hamartoma tumor syndrome: an overview. Genet Med. 2009 Oct;11(10):687-94. doi: 10.1097/GIM.0b013e3181ac9aea. PMID 19668082
- [Background] Usary J, Llaca V, Karaca G, Presswala S, Karaca M, He X, Langerod A, Karesen R, Oh DS, Dressler LG, Lonning PE, Strausberg RL, Chanock S, Borresen-Dale AL, Perou CM. Mutation of GATA3 in human breast tumors. Oncogene. 2004 Oct 7;23(46):7669-78. doi: 10.1038/sj.onc.1207966. PMID 15361840
- [Background] Fararjeh AS, Tu SH, Chen LC, Liu YR, Lin YK, Chang HL, Chang HW, Wu CH, Hwang-Verslues WW, Ho YS. The impact of the effectiveness of GATA3 as a prognostic factor in breast cancer. Hum Pathol. 2018 Oct;80:219-230. doi: 10.1016/j.humpath.2018.06.004. Epub 2018 Jun 11. PMID 29902578
- [Background] Jiang YZ, Yu KD, Zuo WJ, Peng WT, Shao ZM. GATA3 mutations define a unique subtype of luminal-like breast cancer with improved survival. Cancer. 2014 May 1;120(9):1329-37. doi: 10.1002/cncr.28566. Epub 2014 Jan 29. PMID 24477928
- [Background] Takaku M, Grimm SA, Roberts JD, Chrysovergis K, Bennett BD, Myers P, Perera L, Tucker CJ, Perou CM, Wade PA. GATA3 zinc finger 2 mutations reprogram the breast cancer transcriptional network. Nat Commun. 2018 Mar 13;9(1):1059. doi: 10.1038/s41467-018-03478-4. PMID 29535312
- [Background] Annunziato S, de Ruiter JR, Henneman L, Brambillasca CS, Lutz C, Vaillant F, Ferrante F, Drenth AP, van der Burg E, Siteur B, van Gerwen B, de Bruijn R, van Miltenburg MH, Huijbers IJ, van de Ven M, Visvader JE, Lindeman GJ, Wessels LFA, Jonkers J. Comparative oncogenomics identifies combinations of driver genes and drug targets in BRCA1-mutated breast cancer. Nat Commun. 2019 Jan 23;10(1):397. doi: 10.1038/s41467-019-08301-2. PMID 30674894
- [Background] Sheridan W, Scott T, Caroline S, Yvonne Z, Vanessa B, David V, Karen G, Stephen C. Breast cancer in young women: have the prognostic implications of breast cancer subtypes changed over time? Breast Cancer Res Treat. 2014 Oct;147(3):617-29. doi: 10.1007/s10549-014-3125-1. Epub 2014 Sep 11. PMID 25209005
- [Background] Alabdulkareem H, Pinchinat T, Khan S, Landers A, Christos P, Simmons R, Moo TA. The impact of molecular subtype on breast cancer recurrence in young women treated with contemporary adjuvant therapy. Breast J. 2018 Mar;24(2):148-153. doi: 10.1111/tbj.12853. Epub 2017 Jul 14. PMID 28707744
- [Background] Sonderstrup IMH, Jensen MB, Ejlertsen B, Eriksen JO, Gerdes AM, Kruse TA, Larsen MJ, Thomassen M, Laenkholm AV. Evaluation of tumor-infiltrating lymphocytes and association with prognosis in BRCA-mutated breast cancer. Acta Oncol. 2019 Mar;58(3):363-370. doi: 10.1080/0284186X.2018.1539239. Epub 2019 Jan 7. PMID 30614364
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Thomas A, Routh ED, Pullikuth A, Jin G, Su J, Chou JW, Hoadley KA, Print C, Knowlton N, Black MA, Demaria S, Wang E, Bedognetti D, Jones WD, Mehta GA, Gatza ML, Perou CM, Page DB, Triozzi P, Miller LD. Tumor mutational burden is a determinant of immune-mediated survival in breast cancer. Oncoimmunology. 2018 Jul 30;7(10):e1490854. doi: 10.1080/2162402X.2018.1490854. eCollection 2018. PMID 30386679
- [Background] Fountzilas G, Giannoulatou E, Alexopoulou Z, Zagouri F, Timotheadou E, Papadopoulou K, Lakis S, Bobos M, Poulios C, Sotiropoulou M, Lyberopoulou A, Gogas H, Pentheroudakis G, Pectasides D, Koutras A, Christodoulou C, Papandreou C, Samantas E, Papakostas P, Kosmidis P, Bafaloukos D, Karanikiotis C, Dimopoulos MA, Kotoula V. TP53 mutations and protein immunopositivity may predict for poor outcome but also for trastuzumab benefit in patients with early breast cancer treated in the adjuvant setting. Oncotarget. 2016 May 31;7(22):32731-53. doi: 10.18632/oncotarget.9022. PMID 27129168
- [Background] Partridge AH, Hughes ME, Warner ET, Ottesen RA, Wong YN, Edge SB, Theriault RL, Blayney DW, Niland JC, Winer EP, Weeks JC, Tamimi RM. Subtype-Dependent Relationship Between Young Age at Diagnosis and Breast Cancer Survival. J Clin Oncol. 2016 Sep 20;34(27):3308-14. doi: 10.1200/JCO.2015.65.8013. Epub 2016 Aug 1. PMID 27480155